CLINICAL TRIAL: NCT04097158
Title: Oxidative Markers and Efficacy in Amyotrophic Lateral Sclerosis (ALS) Phenotypes Treated With Edaravone
Brief Title: Biomarkers in Different Types of Amyotrophic Lateral Sclerosis (ALS) Patients Being Treated With Edaravone
Status: Recruiting | Type: Observational
Sponsor: Loma Linda University (Other)
Collaborators: Temple University (Other); Thomas Jefferson University (Other); University of Southern California (Other); Northwestern University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB#5190061
Record Dates: First submitted 2019-09-18; First posted 2019-09-20 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Spinal Fluid Urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Upper Motor Neuron predominant ALS
  Interventions: Other: Sample Collection
- Lower Motor Neuron predominant ALS
  Interventions: Other: Sample Collection
- Bulbar predominant ALS
  Interventions: Other: Sample Collection
- Generalized ALS
  Interventions: Other: Sample Collection

INTERVENTIONS:
Other: Sample Collection — The investigators will be collecting blood, urine, and spinal fluid samples.

SUMMARY:
This study is being conducted to help the investigators better understand how the new FDA approved medication Edaravone (also known as Radicava) works in subsets of patients with ALS. The investigators are also trying to understand if there are specific ALS patients, with different presentations of ALS, who might benefit most from this medication. Also, the investigators are following specific biomarkers to determine the optimal treatment duration in patients with different forms of ALS

There is no study medication being offered in this trial. Edaravone is prescribed as part of regular care. In this trial we are collecting blood, urine, and spinal fluid samples in ALS patients who are taking Edaravone and ALS patients who are not taking Edaravone to measure certain markers that could indicate why the drug may be working in a specific type of ALS.

ELIGIBILITY:
Inclusion Criteria:

1. Either possible, probable, or definite ALS, predominantly lower motor neuron disease, predominantly upper motor neuron disease, or bulbar
2. With or without cognitive involvement
3. Willing to participate
4. On no experimental treatment
5. Ages 18 - 85
6. No prior exposure to Edaravone (Radicava)
7. On a stable dose of Riluzole for 30 days or off Riluzole
8. Male or female
9. Females of childbearing age must use contraception

Exclusion Criteria:

1. Unstable medical illness
2. Abnormal liver function (>2x ULN)
3. Unlikely to survive for 26 weeks

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Anyone who meets the Inclusion/Exclusion Criteria
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2019-10-08 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Define pharmacodynamic biomarkers of oxidative stress and antioxidant capacity in different ALS/MND phenotypes. | 6 months
  The investigators aim to identify 4 cohorts of patients with distinct ALS/MND phenotypes and measure a panel of pharmacodynamic biomarkers of oxidative stress and antioxidant capacity in the CSF, blood, and urine.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Rosenfeld, PhD, MD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University, Loma Linda, California, United States